CLINICAL TRIAL: NCT05674214
Title: Occurrence of Liveborn Twins With Birth Weight-discordance and Its Relationship to the Adverse Outcomes: a Multicenter Retrospective Study
Brief Title: Birth Weight-discordance in Twins Pregnancy: a Multicenter Retrospective Study
Status: Completed | Type: Observational
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Peking University Third Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); The Third Hospital Of BaoGang Group (Unknown); Lanzhou University Second Hospital (Other); Yan'an University Affiliated Hospital (Other); Xiamen University Women and Children's Hospital (Unknown); Xinxiang Central Hospital (Other); Central Hospital of Xiaogan (Other); Guizhou Medical University Affiliated Hospital (Unknown); Sichuan Jinxin Women and Children's Hospital (Unknown); The First Affiliated Hospital of Shaoyang University (Unknown); First Affiliated Hospital of Jinan University (Other); First Affiliated Hospital of Shantou University Medical College (Other); Second Affiliated Hospital of Shantou University Medical College (Other); The Second People's Hospital of GuangDong Province (Other); Dongguan People's Hospital (Other Government); Dongguan Binhai Bay Central Hospital (Unknown); Zhongshan People's Hospital, Guangdong, China (Other); Huizhou Municipal Central Hospital (Other); Yuebei People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ThirdGuangzhouMU_QL Cui
Record Dates: First submitted 2022-11-30; First posted 2023-01-06 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-01

CONDITIONS: Twin; Pregnancy, Affecting Fetus or Newborn
Keywords: twins; birth weigh-discordant; occurrence; birth outcomes; multi-center study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- birth weight-discordant group: the birth weight difference within twins is greater than 20%
- the birth weight-concordant group: the birth weight difference within twins is less than or equal to 20%

SUMMARY:
The rate of twin pregnancies in China has increased by 50 percent over the past decade and now stands at about 3 percent. This is significantly higher than the European and American countries. There are significant differences in birth weight of some newborns, that is, birth weight-discordance in twin pregnancies (BWDT). BWDT was significantly associated with fetal death, preterm birth, neonatal death, and neonatal complications. Existing studies mainly focus on the perinatal outcomes of mothers and infants with BWDT, or are reported from small samples in developed countries. The investigators are aware of the need to further explore the occurrence of birth weight inconsistency and adverse neonatal outcomes in China with a large sample. Through retrospective study design, the investigators will collect clinical data of live twin births at multiple study sites, investigate the incidence of BWDT, and analyze its adverse outcomes.

DETAILED DESCRIPTION:
The investigators adopted a multicenter retrospective case-control study design and enrolled live twin births delivered from 2018 to 2020 in 22 hospitals in 12 provinces in China. Children with congenital and hereditary diseases, such as inherited metabolic diseases, complex congenital heart disease, and digestive tract malformations, were excluded from the study. The investigators collected the following information: (1) General information: maternal age, year of delivery, number of delivery, mode of conception, mode of delivery, chorionic nature, education level, newborn sex; (2) Maternal risk factors associated with intrauterine development: induced abortion ≥2 times, placental disease, uterine tumor, gestational diabetes mellitus, gestational hypertension disease, intrahepatic cholestasis, connective tissue disease, hypothyroidism, and chorionic amnitis; (3) Infant birth outcome: gestational age, birth weight, birth length, birth head circumference, very low birth weight infants, ultra-low birth weight infants, the Apgar score, whether transferred to neonatology department. (4) Information of hospitalization during the neonatal period: Pulmonary surfactant use, duration of oxygen therapy, neonatal complications (i.e., pulmonary hemorrhage, BPD, NEC, PDA, ROP, PVL, IVH, anemia, infection, etc.), feeding status (i.e., duration of milk opening, duration of full feeding, feeding style and feeding materials at full feeding, Time to recovery of birth weight), and discharge outcome (i.e., total hospitalization cost, length of stay, gestational age corrected for discharge, discharge status, discharge physique).

ELIGIBILITY:
Inclusion Criteria:

live twin births

1. delivered from 2018 to 2020

Exclusion Criteria:

1. congenital and hereditary diseases
2. inherited metabolic diseases
3. complex congenital heart disease
4. digestive tract malformations

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: live twin births
Sampling Method: Non-Probability Sample
Enrollment: 13440 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
birth outcome | 1 day
  gestational age
neonatal complications | 1 month
  the morbidity of pulmonary hemorrhage, BPD, NEC, PDA, ROP, PVL, IVH, anemia, infection, etc

SECONDARY OUTCOMES:
discharge outcome | 3 months
  total hospitalization cost
discharge outcome | 3 months
  length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Bijun Shi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hiersch L, Barrett J, Aviram A, Mei-Dan E, Yoon EW, Zaltz A, Kingdom J, Melamed N. Patterns of discordant growth and adverse neonatal outcomes in twins. Am J Obstet Gynecol. 2021 Aug;225(2):187.e1-187.e14. doi: 10.1016/j.ajog.2021.01.018. Epub 2021 Jan 25. PMID 33508311
- [Result] D'Antonio F, Thilaganathan B, Laoreti A, Khalil A; Southwest Thames Obstetric Research Collaborative (STORK). Birth-weight discordance and neonatal morbidity in twin pregnancy: analysis of STORK multiple pregnancy cohort. Ultrasound Obstet Gynecol. 2018 Nov;52(5):586-592. doi: 10.1002/uog.18916. Epub 2018 Oct 8. PMID 29028139
- [Result] Jahanfar S, Lim K, Oviedo-Joekes E. Stillbirth Associated With Birth Weight Discordance in Twin Gestations. J Obstet Gynaecol Can. 2019 Jan;41(1):52-58. doi: 10.1016/j.jogc.2018.02.017. Epub 2018 Oct 10. PMID 30316716
- [Result] Miller J, Chauhan SP, Abuhamad AZ. Discordant twins: diagnosis, evaluation and management. Am J Obstet Gynecol. 2012 Jan;206(1):10-20. doi: 10.1016/j.ajog.2011.06.075. Epub 2011 Jun 25. PMID 21864822
- [Result] Diaz-Garcia C, Bernard JP, Ville Y, Salomon LJ. Validity of sonographic prediction of fetal weight and weight discordance in twin pregnancies. Prenat Diagn. 2010 Apr;30(4):361-7. doi: 10.1002/pd.2469. PMID 20187000
- [Result] D'Antonio F, Odibo AO, Prefumo F, Khalil A, Buca D, Flacco ME, Liberati M, Manzoli L, Acharya G. Weight discordance and perinatal mortality in twin pregnancy: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2018 Jul;52(1):11-23. doi: 10.1002/uog.18966. PMID 29155475
- [Result] D'Antonio F, Khalil A, Dias T, Thilaganathan B; Southwest Thames Obstetric Research Collaborative (STORK). Weight discordance and perinatal mortality in twins: analysis of the Southwest Thames Obstetric Research Collaborative (STORK) multiple pregnancy cohort. Ultrasound Obstet Gynecol. 2013 Jun;41(6):643-8. doi: 10.1002/uog.12412. Epub 2013 Apr 22. PMID 23355123